CLINICAL TRIAL: NCT06028997
Title: Implementation of Behavioral and Sleep Hygiene Education With Mindfulness Intervention to Improve Sleep Regularity in Adolescents; is There a Relationship With Anxiety, Depression or Chronotype
Brief Title: Behavioral and Sleep Hygiene Education With Mindfulness Intervention to Improve Sleep Regularity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solveig Magnusdottir (Other Government)
Collaborators: Akureyri Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Solveig Magnusdottir, Chief Medical Officer, Akureyri Hospital
Organization: Akureyri Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VSN-23-086
Record Dates: First submitted 2023-08-29; First posted 2023-09-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Sleep; Depression; Anxiety; Chronotype
Keywords: sleep regularity; sleep duration; adolescents; behavioral therapy; sleep hygiene education; mindfulness intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective cohort-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Behavioral: Behavioral and Sleep Hygiene Education with Mindfulness Intervention

INTERVENTIONS:
Behavioral: Behavioral and Sleep Hygiene Education with Mindfulness Intervention — Education about good sleep hygiene practices and behavior advice to improve sleep based on current literature for 10-15 minutes/week followed by 50 minutes of yoga Nidra and breathing excersices

SUMMARY:
Sleep plays a fundamental role in both mental- and physical-health, with good sleep health including adequate duration and quality, appropriate timing, regularity, and absence of sleep disorders. The purpose of this study is to evaluate sleep in adolescent and if brief behavioral and sleep hygiene education with mindfulness intervention improves, sleep timing, sleep duration, sleep quality, anxiety- and depression symptoms.

During adolescence extensive physiological changes happen that make it easier for adolescents to stay up later, that may increase the time it may take them to fall-asleep and developing insomnia symptoms. At the same time psychosocial changes happen, the societal changes in the last decade may even have further amplified late sleep in adolescents, with increase in social media use and evening screen-time. As sleep need is not decreased and with adolescents having to wake up at "socially acceptable times" rather than the endogenous sleep offset time, sleep duration may be shortened causing chronic sleep loss and daytime sleepiness. Insufficient sleep in adolescents may affect their daytime functioning, causing fatigue and memory issues, affect school attendance and academic performance, affect mood, mental- and physical health, cause behavioral dysfunction and has been associated with worse health outcomes, adverse risk behaviors and even increase risk for accidents.This study should advance understanding of sleep in adolescents and if this simple interventions can be effective in improving their sleep and mental health.

DETAILED DESCRIPTION:
The study is a prospective cohort-study implementing a brief behavioral and sleep hygiene education with mindfulness intervention in adolescents starting a junior collage (16 years of age). All first year students are invited to participate and those interested, willing to sign a consent and have a consent from a parent/guardian will be included in the study, except if diagnosed with chronic atrial fibrillation or ventricular trigemini, severe uncontrolled asthma, or other pulmonary diseases, or diagnosed with moderate or severe obstructive sleep apnea (OSA) then will be excluded from participating in the study.

Sleep duration, sleep timing (sleep onset and conclusion to calculate sleep mid-time and social jetlag), sleep quality, sleep efficiency and wake after sleep onset will be measured with objective home sleep test for three (3) week-nights and two (2) weekend-nights. Sleepiness, insomnia symptoms, anxiety, depression and chronotype will be evaluated with subjective questionnaires before starting intervention of behavioral and sleep hygiene education and mindfulness training once weekly. After the 8-week intervention participants sleep will be measured, sleepiness, insomnia, anxiety, depression symptoms will be re-evaluated with the same questionnaires and their knowledge of how sleep curtailments may affect health and quality of life will be tested.

ELIGIBILITY:
Inclusion Criteria:

First year student attending a junior collage in Northern Europe (Akureyri Iceland)

Exclusion Criteria:

1. chronic atrial fibrillation or ventricular trigemini,
2. severe uncontrolled asthma or other pulmonary diseases,
3. moderate and severe obstructive sleep apnea (OSA)

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Chronotype and relationship with sleep duration, anxiety- and depression symptoms | Baseline and week 9
  Chronotype evaluated with validated sleep questionnaire the Morningness-Eveningness Questionnaire (MEQ), a nineteen-item questionnaire to assess the preferred timing of sleep and activity (outcome presented on scale of 31-86 points) to identify early-, intermediate- and evening chronotypes and evaluate if the different chronotype-groups differ in sleep duration (evaluated in hours and minutes)
Chronotype and relationship with anxiety symptoms | Baseline and week 9
  Chronotype evaluated with validated sleep questionnaire the Morningness-Eveningness Questionnaire (MEQ), a nineteen-item questionnaire to assess the preferred timing of sleep and activity (outcome presented on scale of 31-86 points) to identify early-, intermediate- and evening chronotypes and evaluate if they differ in anxiety symptoms when evaluated with the general anxiety disorder scale-7 (GAD-7), a seven item validated questionnaire designed to screen for and access severity of anxiety (based on scores from 0-21)
Chronotype and relationship with depression symptoms | Baseline and week 9
  Chronotype evaluated with validated sleep questionnaire the Morningness-Eveningness Questionnaire (MEQ), a nineteen-item questionnaire to assess the preferred timing of sleep and activity (outcome presented on scale of 31-86 points) to identify early-, intermediate- and evening chronotypes and evaluate if they differ in depression symptoms when evaluated with the patient health questionnaire (PHQ-9), a nine-item validated questionnaire (scores from 0-27), with higher scores indicating more symptoms
Chronotype and relationship with depression symptoms | Baseline and week 9
  Chronotype evaluated with validated sleep questionnaire the Morningness-Eveningness Questionnaire (MEQ), a nineteen-item questionnaire to assess the preferred timing of sleep and activity (outcome presented on scale of 31-86 points) to identify early-, intermediate- and evening chronotypes and evaluate if they differ in depression symptoms when evaluated with the Becks depression inventory (BDI-II) a ten-item questionnaires to screen for and access severity of depression (scores from 0-63) symptoms, with higher scores indicating more symptoms
Change in sleep regularity and social jetlag from baseline to follow up after 8-weeks of intervention | Baseline and week 9
  Sleep duration, sleep onset and sleep conclusions (all measured in hours and minutes) to calculate sleep midpoint on school- and free days, to calculate social jetlag (in hours and minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Magnusdottir, MD, MSc, MBA, Principal Investigator — MyCardio SleepImage
Locations (2):
- Iceland (2):
  - Menntaskolinn a Akureyri, Akureyri
  - Sjukrahusid a Akureyri, Akureyri

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared